### NCT05175170

## Fertility Decision-Making in Youth and Young Adults

Statistical Analysis Plan Date: 11/7/2022

# Fertility Decision-Making in Youth and Young Adults Statistical Analysis Plan

#### **Primary Outcome: Fertility Knowledge**

We tested the significance of fertility knowledge change among transgender youth and young adults (n=10) and among parents (n=10) between same-day pre-AFFRMED and post-AFFRMED scores using paired samples t-tests. We also calculated the mean difference between pre-AFFRMED and post-AFFRMED scores.

#### **Secondary Outcome: Decision Self-Efficacy**

We tested the change in decision self-efficacy among transgender youth and young adults (n=10) and among parents (n=10) between same-day pre-AFFRMED and post-AFFRMED Decision Self-Efficacy scores using paired samples t-tests. We also calculated the mean difference between pre-AFFRMED and post-AFFRMED Decision Self-Efficacy scores.

#### Other Pre-specified Outcomes: Acceptability, Appropriateness, & Feasibility

Descriptive statistics were used to characterize participants' ratings of AFFRMED acceptability, appropriateness, and feasibility using the Acceptability of Intervention Measure, Intervention Appropriateness Measure, and Feasibility of Intervention Measure.